CLINICAL TRIAL: NCT01889446
Title: Pilot Study to Study the Effects of the Food Preservative Calcium Propionate on Postprandial Hormonal and Metabolic Milieu
Brief Title: The Effects of the Food Preservative Propionic Acid in Post-prandial Metabolism
Acronym: Walnut
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Amir Tirosh, MD,PhD, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2013P001197
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Obesity; Insulin Resistance; Diabetes
Keywords: Propionic acid; Food preservatives
MeSH Terms: conditions — Obesity; Insulin Resistance; Diabetes Mellitus | interventions — calcium propionate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Calcium propionate (Placebo Comparator): Addition of calcium propionate (PA arm) in a capsule (1000 mg) consumed together with a mixed meal of 500 kCal in the morning following an overnight fast. Blood is taken at baseline and every 30 minutes for 4 hours. This arm is compared to a placebo capsule (following identical protocol). Following a washout period of a week, the arms will be crossed over and the PA arm participants will repeat the same protocol in the 'placebo arm'.
  Interventions: Dietary Supplement: Calcium propionate
- Placebo (Placebo Comparator): Addition of placebo (PA arm) in a capsule consumed together with a mixed meal of 500 kCal in the morning following an overnight fast. Blood is taken at baseline and every 30 minutes for 4 hours. This arm is compared to the PA arm (PA, 1000 mg in a capsule). Following a washout period of a week, the arms will be crossed over and the PA arm participants will repeat the same protocol in the 'placebo arm', and vice versa.

INTERVENTIONS:
Dietary Supplement: Calcium propionate
  Arms: Calcium propionate

SUMMARY:
Propionic acid (PA) is used as a preservative in foods such as cheeses, baked goods, or additive for artificial fruit flavors. The U.S. Environmental Protection Agency considers it safe and therefore, has no limitation on its use. Since PA has been shown before to serve as a substrate for glucose production in the liver, the purpose of this study is to find out if PA intake causes changes in levels of glucose, insulin and other important hormones following a meal.

This research study will compare PA to placebo. The placebo looks exactly like the active substance, but it does not contain any active agent (PA). Placebos are used in research studies to see if the results are due to the study drug or to other reasons.

The investigators plan to have 20 subjects take part in this study at the Brigham and Women's Hospital (BWH).

DETAILED DESCRIPTION:
-To test whether PA, added as food supplement to humans, results in altered post-prandial metabolism. The investigators propose to conduct a double-blind, randomized, placebo controlled, cross-over study in which blood levels of metabolites and hormones will be measured in healthy volunteers following a mixed meal test without or with PA.

Study design:

This is a double-blind, randomized, placebo controlled, cross-over study. Twenty volunteers who meet the inclusion/exclusion criteria will be randomized into two groups, provided with a mixed meal without or with calcium proprionate (also known as E282). A week later, participants will be provided with a mixed meal again, following cross-over of the groups. Blood will be collected at baseline, and every 30 minutes for 4 hours.

Study Subjects:

20 healthy male and female volunteers (ages 18 to 65 years) with a body mass index (BMI) of 20 to <30 Kg/m2.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Good health as evidenced by history and physical exam
* BMI: 20-29.9 kg/m2

Exclusion Criteria:

* Fasting plasma glucose >110 mg/dL
* HbA1c >6.0%
* Significant current illness other than treated hypothyroidism
* BP >135/85 or systolic BP <90 mm Hg
* Hepatic disease (transaminase > 3 times normal)
* Renal impairment (Creatinine clearance <60 ml/min)
* History of drug or alcohol abuse
* Participation in any other concurrent clinical trial
* Pregnant women
* History of food allergies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Post prandial insulin levels | During 4 hours after consumption of a meal

CONTACTS AND LOCATIONS:
Overall Officials: Amir Tirosh, MD PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States